| Division | : | Worldwide Development |
|---|---|---|
| Information Type | : | Reporting and Analysis Plan (RAP) |
| Title | : | Reporting and Analysis Plan for A single centre, 2-period, randomized, open-label Phase 1 study to assess the relative bioavailability of a mesylate salt capsule of GSK3640254 compared to a hydrochloride salt capsule in healthy participants |
| <b>Compound Number</b> | : | GSK3640254 |
| Effective Date | : | 21-NOV-2018 |

# **Description:**

• The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 208131 (QCL118221 01)

# **RAP Author(s):**

| Approver | Date | Approval Method |
|---|---|---|
| Principal Statistician (Infectious Disease,<br>Clinical Statistics) | 21-NOV-2018 | E-Signature |
| Associate Manager (SPDS India, Clinical Programming) | 13-NOV-2018 | Review<br>Confirmation<br>Email |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

| RAP Team Review Confirmations<br>(Method: E-mail) | Date |
|----------------------------------------------------------------|-------------|
| Clinical Development Manager (Infectious Disease, CPSSO) | 14-NOV-2018 |
| Physician Product Lead (Clinical Development, ViiV Healthcare) | 13-NOV-2018 |
| Director (Clinical Pharmacology Modelling and Simulation) | 14-NOV-2018 |
| Principal Data Manager (Infectious Disease, Data Management) | 13-NOV-2018 |

# **Clinical Statistics and Clinical Programming Line Approvals:**

# (Method: Pharma TMF eSignature)

| Approver | Date |
|---|---|
| PPD | |
| Statistics Leader (Infectious Disease, Clinical Statistics) On behalf of PPD (Infectious Disease, Senior | 21-NOV-2018 |
| Statistics Director) | |
| Biostatistics and Programming Manager (SPDS India, Clinical Programming) | 21-NOV-2018 |

# **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| 1. | INTRO | ODUCTION | 6 |
| 2. | SLIMA | MARY OF KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | Changes to the Protocol Defined Statistical Analysis Plan | |
| | 2.1. | | |
| | 2.2. | Study Objective(s) and Endpoint(s) | |
| | 2.3.<br>2.4. | Study Design | |
| | 2.4. | Statistical Analyses | / |
| 3. | PLAN | NED ANALYSES | 8 |
| | 3.1. | Interim Analyses | 8 |
| | 3.2. | Final Analyses | 8 |
| 4. | ANAL | YSIS POPULATIONS | 8 |
| | 4.1. | Protocol Deviations | 9 |
| 5. | CONS | SIDERATIONS FOR DATA ANALYSES AND DATA HANDLING | |
| - | | /ENTIONS | 10 |
| | 5.1. | Study Treatment & Sub-group Display Descriptors | 10 |
| | 5.2. | Baseline Definitions | 10 |
| | 5.3. | Multicentre Studies | |
| | 5.4. | Examination of Covariates, Other Strata and Subgroups | |
| | • | 5.4.1. Covariates and Other Strata | |
| | | 5.4.2. Examination of Subgroups | |
| | 5.5. | Multiple Comparisons and Multiplicity | |
| | 5.6. | Other Considerations for Data Analyses and Data Handling | |
| | | Conventions | 11 |
| 6. | STUD | Y POPULATION ANALYSES | 12 |
| | 6.1. | Overview of Planned Study Population Analyses | |
| _ | | , , | |
| 7. | EFFIC | CACY ANALYSES | 12 |
| 8. | SAFE | TY ANALYSES | 12 |
| _ | | Adverse Events Analyses | |
| | 8.2. | Adverse Events of Special Interest Analyses | |
| | 8.3. | Clinical Laboratory Analyses | |
| | 8.4. | Other Safety Analyses | |
| 9. | PΗΔR | RMACOKINETIC ANALYSES | 13 |
| ٥. | 9.1. | Primary Pharmacokinetic Analyses | |
| | 5.1. | 9.1.1. Endpoint / Variables | |
| | | 9.1.1.1. Drug Concentration Measures | |
| | | 9.1.1.2. Derived Pharmacokinetic Parameters | |
| | | 9.1.2. Summary Measure | |
| | | 9.1.3. Population of Interest | |
| | | 9.1.4. Strategy for Intercurrent (Post-Randomization) Events | |
| | | 9.1.5. Statistical Analyses / Methods | |
| | | 9.1.5.1. Statistical Methodology Specification | |
| | | J. I.J. I. Glatistical Mcthodology Openiidation | |

### CONFIDENTIAL

| വ | 80 | 1 | 2 | 4 |
|---|----|---|---|---|
| | υc | ) | J | ш |

| | 9.2.<br>9.3. | | ry Pharmacokinetic Analysespry Pharmacokinetic Analyses | |
|---|---|---|---|---|
| | | - | | |
| 10. | POPU | LATION P | PHARMACOKINETIC (POPPK) ANALYSES | 16 |
| 11. | PHARI | MACODY | NAMIC ANALYSES | 16 |
| 12. | PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES16 | | | |
| 13 | REFE | RENCES | | 17 |
| 14. | | | | 18 |
| | 14.1. | | 1: Protocol Deviation Management and Definitions for Per | 4.0 |
| | | | Population | |
| | 440 | | Exclusions from Per Protocol Population | |
| | 14.2. | | 2: Schedule of Activities | |
| | 440 | | | |
| | 14.3. | | 3: Assessment Windows | |
| | 44.4 | | Definitions of Assessment Windows for Analyses | 22 |
| | 14.4. | | 4: Study Phases and Treatment Emergent Adverse | 00 |
| | | | 0. 1. D | |
| | | 14.4.1. | Study Phases | |
| | | 44.40 | 14.4.1.1. Study Phases for Concomitant Medication | |
| | | 14.4.2. | Treatment Emergent Flag for Adverse Events | |
| | | 14.4.3. | Adverse Events Assignment to Treatment Period | |
| | 115 | 14.4.4. | Concomitant Medication Assignment to Treatment Period | |
| | 14.5. | | 5: Data Display Standards & Handling Conventions | |
| | | 14.5.1. | Reporting Process | |
| | | 14.5.2.<br>14.5.3. | Reporting Standards for Pharmacellinetic | |
| | 14.6. | | Reporting Standards for Pharmacokinetic | |
| | 14.0. | 14.6.1. | General | |
| | | 14.6.1. | | |
| | | 14.6.2.<br>14.6.3. | Study Population | |
| | | 14.6.3. | EfficacySafety | |
| | | 14.6.4.<br>14 6 5 | Pharmacokinetic | |
| | | | Population Pharmacokinetic (PopPK) | |
| | | 14.6.7. | Pharmacodynamic | |
| | 14.7. | | 7: Reporting Standards for Missing Data | 29 |
| | 14.7. | 14.7.1. | Premature Withdrawals | 30 |
| | | 14.7.1. | Handling of Missing Data | |
| | | 14.7.2. | 14.7.2.1. Handling of Missing and Partial Dates | |
| | 14.8. | Annendiy | र 8: Values of Potential Clinical Importance | |
| | 17.0. | 14.8.1. | Laboratory Values | |
| | | 14.8.2. | ECG | |
| | | 14.8.3. | Vital Signs | |
| | | 14.8.4. | Urinalysis | |
| | 14.9. | | s 9: Population Pharmacokinetic (PopPK) Analyses | |
| | 1 1.0. | 14.9.1. | Population Pharmacokinetic (PopPK) Dataset | |
| | | | Specification | 34 |
| | | 14.9.2. | Population Pharmacokinetic (PopPK) Methodology | |
| | 14 10 | | (10: Pharmacokinetic / Pharmacodynamic Analyses | |

### CONFIDENTIAL

| | 14.10.1. | Pharmacokinetic / Pharmacodynamic Dataset | |
|--------|----------|-----------------------------------------------|----|
| | | Specification | |
| | 14.10.2. | Pharmacokinetic / Pharmacodynamic Methodology | 35 |
| 14.11. | Appendix | 11: Abbreviations & Trade Marks | 36 |
| | 14.11.1. | Abbreviations | 36 |
| | | Trademarks | |
| 14.12. | | List of Data Displays | |
| | | Data Display Numbering | |
| | | Mock Example Shell Referencing | |
| | 14.12.3. | Deliverables | 38 |
| | | Study Population Tables | |
| | | Efficacy Tables | |
| | | Efficacy Figures | |
| | | Safety Tables | |
| | | Safety Figures | |
| | | Pharmacokinetic Tables | |
| | | .Pharmacokinetic Figures | |
| | | .Pharmacokinetic Population (PopPK) Tables | |
| | | .Pharmacokinetic Population (PopPK) Figures | |
| | | .Pharmacodynamic Tables | |
| | | .Pharmacodynamic Figures | |
| | | .Pharmacokinetic / Pharmacodynamic Tables | |
| | | .Pharmacokinetic / Pharmacodynamic Figures | |
| | | .ICH Listings | |
| | | .Non-ICH Listings | |
| 14.13. | Appendix | c 13: Example Mock Shells for Data Displays | 51 |

# 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 208131 (QCL118221):

# 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 1 [(Dated: 29/MAY/2018)].

# 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To evaluate the pharmacokinetic (PK) profiles of GSK3640254 following administration of the mesylate salt capsule relative to that of the bishydrochloride salt capsule (reference) in healthy participants | <ul> <li>GSK3640254 area under the curve from time zero to<br/>infinity (AUC<sub>0-∞</sub>), AUC<sub>(0-tlast)</sub>, maximum observed<br/>concentration (C<sub>max</sub>),Time to C<sub>max</sub> (T<sub>max</sub>), Concentration at<br/>24 hours post-dose (C<sub>24h</sub>), relative bioavailability (F<sub>rel</sub>)<br/>based on AUC and C<sub>max</sub></li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To provide additional information of<br>the safety and tolerability of single<br>doses of GSK3640254 in healthy<br>participants | AEs, clinical laboratory values, vital signs,<br>electrocardiogram (ECG) and/or other safety biomarkers |

### 2.3. Study Design

Figure 1 Overview of Study Design



| Overview of S | Study Design and Key Features |
|---|---|
| Design<br>Features | <ul> <li>This is a single centre open-label 2 period cross over study to evaluate the relative bioavailability of a test GSK3640254 mesylate salt capsule against the reference GSK3640254 hydrochloride (HCl) capsule.</li> <li>Each dose of study treatment will be separated by washout period of at least 7 days.</li> </ul> |
| Dosing | <ul> <li>Participants will receive a single 200 mg dose (achieved as 2 x 100 mg capsules) of assigned study treatment during each inpatient period</li> <li>All participants will be dosed in a fed state following a moderate fat meal (approximately 600 calories with approximately 30% of the calories from fat)</li> </ul> |
| Time & Events | Refer to Appendix 2: Schedule of Activities |
| Treatment<br>Assignment | <ul> <li>A randomization schedule was produced using RANDALL NG and distributed to the site pharmacist</li> <li>The randomization number will determine the allocation of treatment sequences (AB or BA)</li> </ul> |
| Interim<br>Analysis | No formal interim analyses are planned for this study. |

# 2.4. Statistical Analyses

No formal statistical hypotheses will be tested. All analyses will be descriptive and exploratory. An estimation approach providing point estimates and corresponding confidence intervals will be used, where appropriate.

### **Relative Bioavailability**

This study is designed to estimate the relative bioavailability of a test GSK3640254 mesylate salt capsule formulation versus the reference HCl capsule formulation. No formal hypothesis will be tested. Separate mixed effects models will be used to analyse the two PK parameters of interest (AUC( $0-\infty$ ) and Cmax). The dependent variable in each model will be the log-transformed PK parameter of interest and the independent variables

will include fixed effects for treatment (mesylate salt capsule or HCl capsule) and period, as well as a random effect for participant. For each primary pharmacokinetic endpoint, point estimates and corresponding 90% confidence intervals will be constructed for the ratio of the geometric mean of the test mesylate salt capsule to the geometric mean of the reference HCl capsule,  $\mu(\text{test})/\mu(\text{reference})$ . More detail is provided in Section 9.1.5.

### 3. PLANNED ANALYSES

## 3.1. Interim Analyses

No formal interim analyses are planned for this study.

### 3.2. Final Analyses

The final planned analyses will be performed after the completion of the following sequential steps:

- 1. All participants have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release (DBR) and database freeze (DBF) has been declared by Data Management.
- 3. All criteria for unblinding the randomization codes have been met.
- 4. Randomization codes have been distributed according to RandAll NG and Quotient procedures.

### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Screened | All participants who were screened for eligibility | Study Population |
| Enrolled | All participants who passed screening and entered the study. Note screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | Study Population |
| Safety | All randomized participants who received at least one dose of study treatment. Participants will be analysed according to the treatment they actually received. | Safety and Study population |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Pharmacokinetic | Participants in the Safety population for whom | PK |
| (PK) | at least one PK sample was obtained, analysed | |
| | and have evaluable drug concentrations | |
| | reported | |

Refer to Appendix 12: List of Data Displays which details the population used for each display.

The "Enrolled" and "Screened" analysis populations were not defined in the study protocol but are defined here to facilitate disclosure requirements and reporting of reasons for screen failure.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan version 1.0 Final dated 24 May 2018.

- Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
- This dataset will be the basis for the summaries and listings of protocol deviations.

A separate summary and/or listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | [RandAll NG] | Data Displays for Reporting | |
| Code | Description | Description | Order in TLF |
| A | An oral dose of 200mg as 2 x GSK3640254 HCl Capsule,100 mg (reference) following a moderate fat meal. | GSK HCI | 1 |
| В | An oral dose of 200 mg as 2 x GSK3640254 Mesylate Salt Capsule, 100 mg (test) following a moderate fat meal. | GSK Mesylate | 2 |

Treatment comparisons will be displayed as follows using the descriptors as specified:

1. GSK3640254 200mg mesylate salt vs GSK3640254 200mg HCl (B vs. A)

### 5.2. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. If time is not collected, Day 1 assessments are assumed to be taken prior to first dose and will be used as baseline. Baseline definitions in the table below are applicable to each period.

| Parameter | Study Asses | Baseline Used in<br>Data Display | | |
|---|---|---|---|---|
| | Screening | Screening Day -1 Day 1 (Pre-Dose) | | |
| Safety | | | | |
| 12-lead ECG | Х | Х | Х | Day 1 (Pre-Dose) |
| Vital Signs | Х | Х | Х | Day 1 (Pre-Dose) |
| Laboratory<br>Assessments | Х | X | | Day -1 |

Unless otherwise stated, if baseline data is missing no derivation will be performed and baseline will be set to missing.

### 5.3. Multicentre Studies

Not applicable.

# 5.4. Examination of Covariates, Other Strata and Subgroups

### 5.4.1. Covariates and Other Strata

Not applicable.

# 5.4.2. Examination of Subgroups

Not applicable.

# 5.5. Multiple Comparisons and Multiplicity

Not applicable.

# 5.6. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

| Section | Component |
|---------|----------------------------------------------------------------|
| 14.3 | Appendix 3: Assessment Windows |
| 14.4 | Appendix 4: Study Phases and Treatment Emergent Adverse Events |
| 14.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 14.6 | Appendix 6: Derived and Transformed Data |
| 14.7 | Appendix 7: Reporting Standards for Missing Data |
| 14.8 | Appendix 8: Values of Potential Clinical Importance |

### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the Safety Population, unless otherwise specified.

Study population analyses including analyses of subject's disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure and treatment compliance will be based on GSK Core Data Standards. Details of the planned displays are presented in Appendix 12: List of Data Displays.

### 7. EFFICACY ANALYSES

Not Applicable.

### 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

### 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 12: List of Data Displays.

## 8.2. Adverse Events of Special Interest Analyses

Not applicable.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Hematology laboratory tests, Urinalysis, and liver function tests will be based on GSK Core Data Standards. The details of the planned displays are in Appendix 12: List of Data Displays.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 12: List of Data Displays.

## 9. PHARMACOKINETIC ANALYSES

## 9.1. Primary Pharmacokinetic Analyses

### 9.1.1. Endpoint / Variables

### 9.1.1.1. Drug Concentration Measures

Pharmacokinetic data will be presented in graphical and/or tabular form and will be summarized descriptively. Plasma GSK3640254 concentration-time data will be listed by participant, treatment group and sampling time and summarized by treatment group and sampling time for each period of the study. Individual participant profiles for GSK3640254 concentration-time data will be presented on both a linear and semi-log scale. Linear and semi-log figures for mean and median GSK3640254 plasma concentrations versus time will also be generated.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 14.5.3 Reporting Standards for Pharmacokinetic)

### 9.1.1.2. Derived Pharmacokinetic Parameters

Derivation of pharmacokinetic parameters will be performed by Quotient under the direct auspices of CPMS, QSci, GlaxoSmithKline. Pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using the currently supported version of WinNonlin. All calculations of non-compartmental parameters will be based on actual sampling times. Pharmacokinetic parameters listed will be determined from the plasma concentration-time data, as data permits.

| Parameter | Parameter Description |
|---|---|
| AUC(0-∞) | Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time. |
| AUC(0-tlast) | Area under the concentration-time curve from time zero to the time of last sample taken |
| C <sub>max</sub> | Maximum observed plasma concentration |
| T <sub>max</sub> | Time to C <sub>max</sub> |
| C <sub>24h</sub> | Concentration at 24 hrs post dose |
| C <sub>last</sub> | Observed plasma concentration at T <sub>last</sub> |
| T <sub>last</sub> | Time from dosing at which GSK3640254 was last quantifiable in a concentration vs. time profile |
| T <sub>lag</sub> | The elapsed time from dosing at which GSK3640254 was first quantifiable in a concentration vs time profile. |

| Parameter | Parameter Description |
|---|---|
| AUC <sub>%Extrap</sub> | The percentage of AUC extrapolated beyond the last measured time point |
| t½ | Apparent terminal phase half-life, calculated as; t½ = ln2 / lambda_z |
| Vd/F | The apparent volume of distribution following extravascular dosing |
| CI/F | Oral clearance, the apparent volume of plasma cleared of GSK3640254 per unit time following extravascular dosing. |
| Lambdaz | Terminal phase rate constant |

#### NOTES:

Additional parameters may be included as required.

All the derived parameters described above will be listed. For each of these parameters, except tmax and tlag, the following summary statistics will be calculated for each treatment group: n, arithmetic mean, standard deviation (SD), median, minimum, maximum, geometric mean with associated 95% CI, standard deviation of logarithmically transformed data, and the between-participant CV (%CVb) (where %CVb =  $100*\sqrt{\exp(SD^2)-1}$ ) based on the geometric mean for the log-transformed PK parameters. For tmax and tlag, median, maximum, minimum, arithmetic mean and standard deviation will be calculated.

### 9.1.2. Summary Measure

The parameters used for the treatment comparison of relative bioavailability of the single dose of the mesylate salt capsule relative to the single dose of the HCl capsule will be area under concentration time curve (AUC(0- $\infty$ ) or AUC(0-tlast) if AUC(0- $\infty$ ) cannot be derived) and  $C_{max}$ .

### 9.1.3. Population of Interest

The primary pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

### 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

Not applicable.

## 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 12: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

### 9.1.5.1. Statistical Methodology Specification

The following pharmacokinetic statistical analyses will only be performed if sufficient data is available (i.e. if participants have well defined plasma profiles).

### **Endpoint / Variables**

AUC(0-∞) (or AUC(0-tlast) if AUC(0-∞) cannot be derived) and Cmax

### **Model Specification**

AUC(0-∞) and Cmax will be separately analysed using a mixed effects models. In each model
the dependent variable will be the log-transformed PK parameter of interest (AUC(0-∞) or
Cmax). The independent variables will include fixed effects for treatment (mesylate salt
capsule or HCl capsule) and period, and a random effect for participant.

### **Model Checking & Diagnostics**

- An unstructured covariance structure for the R matrix will be used by specifying "type=un" on the RANDOM line
- In the event that this model fails to converge, alternative correlation structures may be considered such as CSH or CS.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.
- Normality assumptions underlying the model used for analysis will be examined by
  obtaining a normal probability plot of the residuals and a plot of the residuals versus the
  fitted values (i.e. checking the normality assumption and constant variance assumption of
  the model respectively) to gain confidence that the model assumptions are reasonable.
- If there are any departures from the distributional assumptions, alternative models will be explored using appropriate transformed data.

### **Model Results Presentation**

- The estimated difference and CI obtained on the log scale will be exponentiated to provide an estimate of the fed to fasted ratio and its associated 90% CI. Estimates of within-subject variability (%CVw) will also be provided (%CVw=SQRT(exp(MSE) – 1)×100). %CVw represents a pooled measure of within-subject variability across all treatments.
- Comparative plots of individual PK parameters will be generated by treatment on linear and semi-logarithmic scales.
- Plots of adjusted geometric mean ratio of test to reference treatment together with 90% confidence intervals will be produced.
- Listing of individual PK parameter ratios will be generated.
- Supportive SAS output from statistical analysis will be generated.

### Subgroup Analyses

Not Applicable.

### **Sensitivity and Supportive Analyses**

Not Applicable.

# 9.2. Secondary Pharmacokinetic Analyses

Not applicable.

# 9.3. Exploratory Pharmacokinetic Analyses

Not Applicable.

# 10. POPULATION PHARMACOKINETIC (POPPK) ANALYSES

Not Applicable

# 11. PHARMACODYNAMIC ANALYSES

Not applicable.

# 12. PHARMACOKINETIC / PHARMACODYNAMIC ANALYSES

Not applicable.

# 13. REFERENCES

GUI\_51487: Non-compartmental Analysis of Pharmacokinetic Data, CPMS Global. Effective Date: 01-NOV-2017

GlaxoSmithKline Document Number 2017N346490\_01: A single centre, 2-period, randomized, open-label Phase 1 study to assess the relative bioavailability of a mesylate salt capsule of GSK3640254 compared to a hydrochloride salt capsule in healthy participants. Effective Date: 29-MAY-2018

# 14. APPENDICES

# 14.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

These details are documented in the Protocol Deviation Management Plan (PDMP).

# 14.1.1. Exclusions from Per Protocol Population

Not applicable.

# 14.2. Appendix 2: Schedule of Activities

# 14.2.1. Protocol Defined Schedule of Events

Table 1 Schedule of Activities

| Procedure | Screening<br>(up to 28 | | Treat | ment Peri | | Follow-up<br>(7 to 10 days | Notes | | |
|---|---|---|---|---|---|---|---|---|---|
| | days<br>before<br>Day 1) | 1 | 1 | 2 | 3 | 4 | post last dose)<br>or Early<br>Discontinuation | | |
| Outpatient visit | Х | | | | | Х | Х | | |
| Inpatient stay | | X <sup>1</sup> | Х | Х | X <sup>2</sup> | | | 1. | Admission in the morning Furlough from unit after assessment s |
| Informed consent | Х | | | | | | | | |
| Inclusion and exclusion criteria | Х | X3 | | | | | | 3. | Recheck<br>clinical<br>status at<br>admission<br>of Period 1 |
| Demography | Х | | | | | | | | |
| Full physical<br>examination<br>including<br>height and<br>weight <sup>4</sup> | Х | | | | | | | 4. | See<br>protocol<br>Section<br>9.4.1 for<br>systems to<br>be<br>examined |
| Columbia Suicide Severity Rating Scale (CSSRS) | X | | | | X | | | | |
| Brief physical examination | | | <b>X</b> <sup>5</sup> | | <b>X</b> <sup>5</sup> | | X | 5. | Pre-dose<br>and 48 h<br>post-dose<br>See<br>protocol<br>Section<br>9.4.1 for<br>systems to<br>be<br>examined |

| Procedure | Screening<br>(up to 28 | | Treat | ment Perio | | Follow-up<br>(7 to 10 days | Notes | | |
|---|---|---|---|---|---|---|---|---|---|
| | days<br>before<br>Day 1) | 1 | 1 | 2 | 3 | 4 | post last dose)<br>or Early<br>Discontinuation | | |
| Medical history<br>(includes<br>substance<br>usage) <sup>6</sup> | X | | | | | | | | Substances:<br>Drugs,<br>alcohol,<br>tobacco and<br>caffeine |
| Urine pregnancy test <sup>7</sup> | Х | Х | | | | | Х | | All female participants |
| Follicle<br>stimulating<br>hormone<br>(FSH) <sup>8</sup> | Х | | | | | | | | As needed<br>in women to<br>confirm<br>postmenopa<br>usal status |
| HIV, Hepatitis<br>B and C<br>screening | Х | | | | | | | | |
| Urine drug<br>screen | Х | Х | | | | | | | |
| Alcohol breath test | Х | Х | | | | | | | |
| Carbon<br>monoxide<br>breath test | Х | Х | | | | | | | |
| Laboratory<br>assessments<br>(haematology,<br>clinical<br>chemistry and<br>urinalysis) | Х | X9 | | | Xa | | X | | 48 h post-<br>dose<br>Allowable<br>windows in<br>protocol<br>Section<br>9.4.4 |
| 12-lead ECG | Х | Х | X <sup>10</sup> | X <sup>10</sup> | | X <sup>10</sup> | X | | Time points<br>in Table 2<br>Allowable<br>windows in<br>protocol<br>Section<br>9.4.3 |
| Vital signs | Х | Х | X <sup>11</sup> | X11 | | X <sup>11</sup> | X | 11. | Time points<br>in Table 2<br>Allowable<br>windows in<br>protocol<br>Section<br>9.4.2 |

| Procedure | Screening<br>(up to 28 | Treatment | | | ods 1 and | Follow-up<br>(7 to 10 days | Notes | |
|---|---|---|---|---|---|---|---|---|
| | days<br>before<br>Day 1) | 1 | 1 | 2 | 3 | 4 | post last dose)<br>or Early<br>Discontinuation | |
| Randomization | | | X <sup>12</sup> | | | | | 12. Pre-dose<br>Period 1<br>only |
| Study<br>treatment | | | Х | | | | | |
| AE review | | Х | <b>←====</b> | ====== | ====== | =====> | X | |
| SAE review | Х | Х | <b>←====</b> | ====== | ====== | =====> | X | |
| Concomitant medication review | | Х | <b>←===</b> | ====== | ====== | =====> | Х | |
| PK blood<br>sample<br>collection <sup>13</sup> | | | <b>←===</b> = | ====== | ====== | ===== | | 13. Time points in Table 2 |

Table 2 Pharmacokinetic Blood Sampling Collection, ECG ad Vital Sign Times

| | | Treatment Periods 1 and 2 | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time (h) | Pre-<br>dose | 0 | 0.5 | 1 | 1.5 | 2 | 3 | 4 | 5 | 6 | 8 | 12 | 24 | 36 | 48 | 72 |
| Dosing | | Х | | | | | | | | | | | | | | |
| PK<br>Sampling | Х | | Х | Х | Χ | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х |
| Single 12-<br>lead ECG<br>(repeat<br>allowed) | X | | | | | X | | X | | Х | | | Х | | | Х |
| Single set<br>of Vital<br>signs | Х | | | | | X | | X | | Х | | | X | | | Х |

# 14.3. Appendix 3: Assessment Windows

# 14.3.1. Definitions of Assessment Windows for Analyses

All acceptable assessment windows are defined in Section 9.4.2 (vitals), Section 9.4.3 (ECG), Section 9.4.4 (clinical safety laboratory assessments), and Section 9.5 (PK) of the protocol. No assessment windows will be redefined in the RAP.

# 14.4. Appendix 4: Study Phases and Treatment Emergent Adverse Events

### 14.4.1. Study Phases

Assessments and events will be classified according to the time of occurrence relative to administration of study treatment. Study phases are defined separately for each period. Period 1

| <b>Study Phase</b> | Definition |
|---|---|
| Pre-Treatment | Date < Period 1 Study Treatment Start Date/Time |
| On-Treatment | Period 1 Study Treatment Start Date/Time ≤ Date < Period 1 Study Treatment Start Date/Time + 5 days |
| Post-Treatment | Period 1 Study Treatment Start Date/Time + 5 days < Date |

### Period 2

| Study Phase | Definition |
|---|---|
| Pre-Treatment | Date < Period 1 Study Treatment Start Date/Time |
| On-Treatment | Period 2 Study Treatment Start Date/Time ≤ Date < Period 2 Study Treatment Start Date/Time + 5 days |
| Post-Treatment | Period 2 Study Treatment Start Date/Time + 5 days < Date |

### 14.4.1.1. Study Phases for Concomitant Medication

| Study Phase | Definition |
|---|---|
| Prior | If medication end date is not missing and is prior to screening visit |
| Concomitant | Any medication that is not a prior |

### NOTES:

 Please refer to Appendix 7: Reporting Standards for Missing Data for handling of missing and partial dates for concomitant medication. Use the rules in this table if concomitant medication date is completely missing.

### 14.4.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment<br>Emergent | <ul> <li>If AE onset date is on or after treatment start date &amp; on or before treatment stop date. (plus washout or protocol-specified time limit (e.g. half-life of drug, certain number of days, etc.).</li> <li>Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date</li> </ul> |
| | <ul> <li>For studies with greater than one treatment period (e.g., crossover study), if AE onset is during one period and worsens during a later period it would be counted in both periods. For the initial period the logic would be as above. For the later period the logic would use the treatment dates associated with the later period:</li> <li>Treatment Period Start Date ≤ AE Worsening Date ≤ Study Treatment Stop Date</li> </ul> |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

### 14.4.3. Adverse Events Assignment to Treatment Period

Adverse events (AEs) will be assigned to a treatment period and corresponding treatment received in that treatment period after the imputations defined in RAP Section 14.7.2.1 have been performed.

- Treatment Period 1: all AEs with start date/time at the time of or after IMP administration in Treatment Period 1 and before IMP administration in Treatment Period 2
- Treatment Period 2: all AEs with start date/time at the time of or after IMP administration in Treatment Period 2

Thus, AEs occurring during the 1<sup>st</sup> washout will be assigned to the treatment received in Treatment Period 1 and AEs occurring during follow-up will be assigned to the treatment received in Treatment Period 2.

### 14.4.4. Concomitant Medication Assignment to Treatment Period

Concomitant medications (CMs) will be assigned to a treatment period and corresponding treatment received in that treatment period after the imputations defined in RAP Section 14.7.2.1 have been performed.

- Treatment Period 1: all CMs with start date/time at the time of or after IMP administration in Treatment Period 1 and before IMP administration in Treatment Period 2
- Treatment Period 2: all CMs with start date/time at the time of or after IMP administration in Treatment Period 2

Thus, CMs occurring during the washout period will be assigned to the treatment received in Treatment Period 1, and CMs occurring during follow-up will be assigned to the treatment received in Treatment Period 2.

# 14.5. Appendix 5: Data Display Standards & Handling Conventions

## 14.5.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS and WinNonLin software will be used. | |
| Reporting Area | |
| HARP Server | : \\us1salx00259.corpnet2.com |
| HARP Compound | HARP Compound : \arwork\gsk3640254\mid208121\final_01 |
| <b>Analysis Datasets</b> | |
| <ul> <li>Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.2 &amp; ADaM IG<br/>Version 1.0.</li> </ul> | |
| Generation of RTF Files | |
| <ul> <li>RTF files will be generated for Tables, one RTF file per item. Listings will be generated in L10 format, and Figures will be generated in PDF format.</li> </ul> | |

## 14.5.2. Reporting Standards

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:
  - https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics
- Do not include subject level listings in the main body of the GSK Clinical Study Report. All subject level listings should be located in the modular appendices as ICH or non-ICH listings

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| <ul> <li>Unscheduled visits</li> </ul> | <ul> <li>Unscheduled visits will not be included in summary tables and/or figures.</li> </ul> |
| All unscheduled vis | sits will be included in listings. |
| <b>Descriptive Summary</b> | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | ategorical Data N, n, frequency, % |
| Graphical Displays | |
| Refer to IDSL State | tistical Principals 7.01 to 7.13. |
| Note | |
| | All displays (TFL) will use the term "Subjects" in order to reflect GSK Display Standards and CDISC SDTM/ADaM standards). The term "Subjects" is used to refer to the "Participants" in the protocol. |

# 14.5.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Con | centration Data |
|---|---|
| PC Windows Non-<br>Linear (WNL) File | PC WNL file (CSV format) for the non-compartmental analysis by Clinical Pharmacology Modelling and Simulation function will be created according to [Standards for the Transfer and Reporting of PK Data using HARP ("PK One" document)]. Note: Concentration values will be imputed as per GUI_51487 |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. Refer to IDSL Statistical Principle 6.06.1. Note: Concentration values will be imputed as per GUI_51487 for descriptive summary statistics/analysis and summarized graphical displays only. |
| Pharmacokinetic Para | Pharmacokinetic Parameter Derivation |
| PK Parameter to be<br>Derived by<br>Programmer | The following PK parameters will be derived by the Programmer: FRel |
| Pharmacokinetic Para | ameter Data |
| Is NQ impacted PK<br>Parameters Rule<br>Being Followed | Yes, refer to Standards for Handling NQ Impacted PK Parameters |
| Descriptive Summary<br>Statistics, Graphical<br>Displays and Listings | Refer to IDSL PK Display Standards. |

### 14.6. Appendix 6: Derived and Transformed Data

### 14.6.1. General

### **Multiple Measurements at One Analysis Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from First Dose Date:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < First Dose Date → Study Day = Ref Date First Dose Date
  - Ref Data ≥ First Dose Date → Study Day = Ref Date (First Dose Date) + 1

## 14.6.2. Study Population

### **Treatment Compliance**

Treatment compliance will be calculated based on the formula:

# Treatment Compliance = Number of Actual Doses / (Planned Treatment Duration in Days \* Frequency)

- Frequency is 2 for BID and 1 for QD. Treatment compliance could be greater than 100% if there are events of overdose. Cumulative compliance (since Day 1) at each visit will be calculated.
- Planned Treatment Duration is defined as one day.

#### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:

### Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- The cumulative dose will be based on the formula:

### **Cumulative Dose = Sum of (Number of Days x Total Daily Dose)**

If there are any treatment breaks during the study, exposure data will be adjusted accordingly.

### 14.6.3. Efficacy

Not applicable.

### 14.6.4. Safety

### **ECG Parameters**

#### RR Interval

IF RR interval (msec) is not provided directly, then RR can be derived as:

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcF} \right)^3 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Fredericia's (QTcF) formula will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcF and/or QTcB will be derived as:

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

# **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the smallest unit of one more significant digit than the number of significant digits in the observed values will be added or subtracted (whichever is applicable) in order to impute the corresponding number. For example:
  - o Example 1: 2 significant digits (as in "<2.2") will be imputed as 2.19
  - Example 2: 1 significant digit (as in ">5") will be imputed as 5.1
  - Example 3: 0 significant digits (as in "<0") will be imputed as -1".</li>
  - There will be no imputation in the data listings; all values will be displayed as recorded in the database.

### 14.6.5. Pharmacokinetic

Calculation of Pharmacokinetic Parameter Values Not Described in Section 9 (refer to GUI\_51487 for pharmacokinetic analysis information)

### lambda\_z (terminal phase rate constant)

• Slope of the line determined by linear regression of logarithmically transformed concentration v. time data

# %AUCex (percentage of AUC(0-∞) obtained by extrapolation)

• Calculated as 100 x [AUC(0-∞) – AUC(0-tlast)] / AUC(0-∞)

# 14.6.6. Population Pharmacokinetic (PopPK)

Not applicable.

# 14.6.7. Pharmacodynamic

Not applicable.

# 14.7. Appendix 7: Reporting Standards for Missing Data

# 14.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as if he/she completed all periods of the study including the last scheduled follow-up visit</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>Withdrawal visits will be slotted as per Appendix 3: Assessment Windows or will be summarised as withdrawal visits.</li> </ul> |

# 14.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: |
| | <ul> <li>These data will be indicated by the use of a "blank" in subject listing displays.</li> <li>Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be<br/>missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 14.7.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |
| Concomitant<br>Medications/<br>Medical<br>History | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 14.8. Appendix 8: Values of Potential Clinical Importance

# 14.8.1. Laboratory Values

Division of AIDS (DAIDS, Version 2.0, November 2014) AE grades 2, 3, and 4 of lab abnormalities will be listed by subject, period/treatment, visit, and actual date and time.

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Potential Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | D-#f | Male | | 0.54 |
| Hematocrit | Ratio of | Female | | 0.54 |
| | I | $\Delta$ from BL | ↓0.075 | |
| | /1 | Male | | 180 |
| Haemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x10 <sup>9</sup> / L | | 0.8 | |
| Neutrophil Count | x10 <sup>9</sup> / L | | 1.5 | |
| Platelet Count | x10 <sup>9</sup> / L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 12 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Potential Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Bicarbonates | mmol/L | | 18 | 32 |
| BUN | mmol/L | | | >9 |
| Calcium | mmol/L | | 2 | 2.75 |
| Chloride | mmol/L | | 98 | 107 |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ <b>44.2</b> |
| Glucose (fasting) | mmol/L | | 3 | 9 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total Protein | g/L | $\Delta$ from BL | < -15 | >15 |

| Liver Function | | | |
|---|---|---|---|
| Test Analyte | Units | Category | Potential Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| Alkaline phosphatase | U/L | High | ≥ 2x ULN |
| Total Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| Total Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

### 14.8.2. ECG

| ECG Parameter | Units | Potential Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| PR Interval | msec | <120 | >200 |
| QRS Interval | msec | < 60 | >120 |
| QTcF Interval | msec | < 320 | >450 |
| RR Interval | msec | < 600 | > 1200 |
| Change from Baseline | | | |
| Increase from Baseline QTc | msec | | >60 |

# 14.8.3. Vital Signs

| Vital Sign Parameter | Units | Potential Clinical Concern Range | |
|---|---|---|---|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | <85 | >140 |
| Diastolic Blood Pressure | mmHg | <45 | >90 |
| Heart Rate | bpm | <40 | >100 |
| Respiratory Rate | Breaths/min | 12 | 20 |

# 14.8.4. Urinalysis

Per IDSL standards, a subject is considered to have urinalysis results of PCI, if there is an increase in Protein or an increase in Occult Blood results during the study, or if microscopy is performed.

- 14.9. Appendix 9: Population Pharmacokinetic (PopPK) Analyses
- **14.9.1.** Population Pharmacokinetic (PopPK) Dataset Specification Not applicable.
- **14.9.2.** Population Pharmacokinetic (PopPK) Methodology Not applicable.

- 14.10. Appendix 10: Pharmacokinetic / Pharmacodynamic Analyses
- 14.10.1. Pharmacokinetic / Pharmacodynamic Dataset Specification

Not applicable.

14.10.2. Pharmacokinetic / Pharmacodynamic Methodology

Not applicable.

# 14.11. Appendix 11: Abbreviations & Trade Marks

# 14.11.1. Abbreviations

| Abbreviation Description ADaM Analysis Data Model AE Adverse Event AIC Akaike's Information Criteria ALT Alanine Aminotransferase AST Aspartate Aminotransferase A&R Analysis and Reporting CDISC Clinical Data Interchange Standards Consortium |
|---|
| AE Adverse Event AIC Akaike's Information Criteria ALT Alanine Aminotransferase AST Aspartate Aminotransferase A&R Analysis and Reporting CDISC Clinical Data Interchange Standards Consortium |
| AIC Akaike's Information Criteria ALT Alanine Aminotransferase AST Aspartate Aminotransferase A&R Analysis and Reporting CDISC Clinical Data Interchange Standards Consortium |
| ALT Alanine Aminotransferase AST Aspartate Aminotransferase A&R Analysis and Reporting CDISC Clinical Data Interchange Standards Consortium |
| AST Aspartate Aminotransferase A&R Analysis and Reporting CDISC Clinical Data Interchange Standards Consortium |
| A&R Analysis and Reporting CDISC Clinical Data Interchange Standards Consortium |
| CDISC Clinical Data Interchange Standards Consortium |
| <b>U</b> |
| CI Confidence Interval |
| CPMS Clinical Pharmacology Modelling & Simulation CS Clinical Statistics |
| CSR Clinical Study Report |
| CTR Clinical Trial Register |
| CV <sub>b</sub> / CV <sub>w</sub> Coefficient of Variation (Between) / Coefficient of Variation (Within) |
| DBF Database Freeze |
| DBR Database Release |
| DOB Date of Birth |
| DP Decimal Places |
| eCRF Electronic Case Record Form |
| EMA European Medicines Agency |
| FDA Food and Drug Administration |
| FDAAA Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK GlaxoSmithKline |
| IA Interim Analysis |
| ICH International Conference on Harmonization |
| IDMC Independent Data Monitoring Committee |
| IDSL Integrated Data Standards Library |
| IMMS International Modules Management System |
| IP Investigational Product |
| ITT Intent-To-Treat |
| MMRM Mixed Model Repeated Measures |
| PCI Potential Clinical Importance |
| PD Pharmacodynamic |
| PDMP Protocol Deviation Management Plan |
| PK Pharmacokinetic |
| PP Per Protocol |
| PopPK Population PK |
| QC Quality Control |
| QTcF Frederica's QT Interval Corrected for Heart Rate |
| QTcB Bazett's QT Interval Corrected for Heart Rate |
| RAP Reporting & Analysis Plan |
| RAMOS Randomization & Medication Ordering System |
| Abbreviation | Description |
|--------------|-----------------------------------------|
| SAC | Statistical Analysis Complete |
| SDSP | Study Data Standardization Plan |
| SDTM | Study Data Tabulation Model |
| SGOT | Serum Glutamic-Oxaloacetic Transaminase |
| SGPT | Serum Glutamic-Pyruvic Transaminase |
| SOP | Standard Operation Procedure |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

### 14.11.2. Trademarks

| Trademarks of the GlaxoSmithKline Group of Companies |
|------------------------------------------------------|
| NONE |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Phoenix |
| SAS |
| WinNonlin |

#### 14.12. Appendix 12: List of Data Displays

#### 14.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------------------------|----------------|----------------|
| Study Population | 1.1 to 1.12 | Not applicable |
| Efficacy | Not applicable | Not applicable |
| Safety | 3.1 to 3.18 | 3.1 to 3.3 |
| Pharmacokinetic | 4.1 to 4.7 | 4.1 to 4.5 |
| Population Pharmacokinetic (PopPK) | Not applicable | Not applicable |
| Pharmacodynamic and / or Biomarker | Not applicable | Not applicable |
| Pharmacokinetic / Pharmacodynamic | Not applicable | Not applicable |
| Section | List | ings |
| ICH Listings | 1 to | 35 |
| Other Listings | 3 | 6 |

#### 14.12.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 13: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 14.12.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [1] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 14.12.4. Study Population Tables

| Study F | opulation Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition | | | | |
| 1.1. | Safety | ES1A | Summary of Participant Disposition for the Participant Conclusion Record | ICH E3, FDAAA, EudraCT | SAC [1] |
| 1.2. | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC [1] |
| 1.3. | Safety | ES4 | Summary of Participant Disposition at Each Study Epoch | ICH E3 | SAC [1] |
| 1.4. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements | SAC [1] |
| 1.5. | Enrolled | NS1 | Summary of Number of Participant by Country and Site ID | EudraCT/Clinical Operations. For crossover studies, only a total column should be used; the number of subjects will not be broken down by treatment group. | SAC [1] |
| Protoco | ol Deviation | | | | |
| 1.6. | Safety | DV1 | Summary of Important Protocol Deviations | ICH E3. Only total column is needed since this is a crossover study. | SAC [1] |
| Populat | tion Analysed | | | | |
| 1.7. | Screened | SP1 | Summary of Study Populations | IDSL | SAC [1] |

| Study F | Population Tab | les | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.8. | Safety | DM3 | Summary of Demographic Characteristics | ICH E3, FDAAA, EudraCT | SAC [1] |
| 1.9. | Enrolled | DM11 | Summary of Age Ranges | EudraCT, Only include total column | SAC [1] |
| 1.10. | Safety | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT, Only include total column | SAC [1] |
| Prior a | nd Concomitan | t Medications | | | |
| 1.11. | Safety | MH4 | Summary of Medical Conditions | ICH E3 | SAC [1] |
| 1.12. | Safety | CM1 | Summary of Concomitant Medications | ICH E3 | SAC [1] |

## 14.12.5. Efficacy Tables

Not applicable.

## 14.12.6. Efficacy Figures

Not applicable.

# 14.12.7. Safety Tables

| Tables | | | | |
|---|---|---|---|---|
| Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| e Events (AEs) | | | | |
| Safety | AE5A | Summary of All Adverse Events by Maximum Intensity by System Organ Class and Preferred Term | ICH E3, Include column for total across all intensities | SAC [1] |
| Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency | ICH E3 | SAC [1] |
| Safety | AE5A | Summary of All Drug-Related Adverse Events by System Organ Class and Preferred Term and Maximum Intensity | ICH E3 | SAC [1] |
| Safety | AE15 | Summary of Non-serious Adverse Events by System Organ Class and Preferred Term (Number of Participant and Occurrences) | FDAAA, EudraCT | SAC [1] |
| tory: Chemistry | / | | | |
| Safety | LB1 | Summary of Clinical Chemistry Changes from Baseline | ICH E3 | SAC [1] |
| tory: Hematolo | gy | | | |
| Safety | LB1 | Summary of Hematology Changes from Baseline | ICH E3 | SAC [1] |
| Safety | LB17 | Summary of Worst Case Hematology Results by PCI Criteria Post-Baseline Relative to Baseline | ICH E3 | SAC [1] |
| tory: Urinalysis | <b>.</b> | | | |
| Safety | UR1 | Summary of All Urinalysis Results by Visit | | SAC [1] |
| tory: Hepatobil | iary (Liver) | | | |
| Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | IDSL | SAC [1] |
| | Safety Safety Safety Safety Safety tory: Chemistry Safety Safety tory: Hematolo Safety Safety Safety tory: Urinalysis Safety tory: Hepatobil | Population IDSL / Example Shell e Events (AEs) Safety AE5A Safety AE5A Safety AE15 tory: Chemistry Safety LB1 tory: Hematology Safety LB1 Safety LB1 tory: Urinalysis Safety UR1 tory: Hepatobiliary (Liver) | Population IDSL / Example Shell Title | Population DSL / Example Shell Title Programming Notes |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| ECG | | | | | |
| 3.10. | Safety | EG1 | Summary of ECG Findings | IDSL | SAC [1] |
| 3.11. | Safety | EG10 | Summary of Maximum QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC [1] |
| 3.12. | Safety | Table 10.17<br>from Study<br>HAI115711 | Summary of Category of QTc Data by Treatment and Visit | | SAC [1] |
| 3.13. | Safety | EG11 | Summary of Maximum Increase in QTc Values Post-Baseline Relative to Baseline by Category | IDSL | SAC [1] |
| 3.14. | Safety | Table 10.18<br>from Study<br>HAI115711 | Summary of Category of QTc Change from Baseline by Treatment and Visit | | SAC [1] |
| 3.15. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | IDSL, Include Baseline values | SAC [1] |
| Vital Si | gns | | | | • |
| 3.16. | Safety | VS1 | Summary of Vital Signs | ICH E3 | SAC [1] |
| 3.17. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | ICH E3 | SAC [1] |
| Other | | | | | |
| 3.18. | Safety | CSSRS4 | Listing of C-SSRS Suicidal Ideation or Behaviour Data | IDSL | SAC [1] |

## 14.12.8. Safety Figures

| Safety: | Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Laborat | tory | | | | |
| 3.1. | Safety | As EG9 | Line Plot of Selected Clinical Lab Tests Mean (95% CI) Change from Baseline by Treatment and Time | Only include scheduled visits and for selected lab test (ALT, AST, Bili) Plots will be presented with treatment groups overlaid | SAC [1] |
| ECG | | | | | |
| 3.2. | Safety | EG9 | Line Plot of Mean (95% CI) Change from Baseline of ECG Data by Treatment and Time | Plots will be presented with treatment groups overlaid | SAC [1] |
| | | | | Include plots on separate pages for QT, QTcF, QTcB, PR, and QRS | |
| Vital Sig | gns | | | | |
| 3.3. | Safety | As EG9 | Line Plot of Mean (95% CI) Change from Baseline for Vital Signs by Treatment and Time | Plots will be presented with treatment groups overlaid | SAC [1] |
| | ļ | | | Include plots on separate pages for SBP, DBP, HR | |

#### 14.12.9. Pharmacokinetic Tables

| Pharma | Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Bioava | ilability | | | | |
| 4.1. | PK | PK01 | Summary of Plasma GSK3640254 Pharmacokinetic Concentration-Time Data by Treatment | | SAC [1] |
| 4.2. | PK | PK04 | Summary of Derived Plasma GSK3640254 Pharmacokinetic Parameters by Treatment | | SAC [1] |
| 4.3. | PK | PK05 | Summary Statistics of Log-Transformed Derived Plasma GSK3640254 Pharmacokinetic Parameters by treatment | | SAC [1] |
| 4.4. | PK | Non-Standard1 | Summary of Result of Plasma GSK3640254 Pharmacokinetic Parameter Treatment Comparisons for Relative Bioavailability | PK Parameters: AUC(0-inf), and Cmax Ratio: Test/Reference (Mesylate/HCI) | SAC [1] |
| 4.5. | PK | PK14 | Listing of Derived Plasma GSK3640254 Pharmacokinetic Parameters by treatment | Sort by participant and treatment | SAC [1] |
| 4.6. | PK | PK08 | Listing of Plasma GSK3640254 Pharmacokinetic Concentration-<br>Time Data by treatment | Sort by participant, period, day, and time | SAC [1] |
| 4.7. | PK | PK15 | Listing of Individual Derived Plasma GSK3640254 Pharmacokinetic Parameters Treatment Ratios | PK Parameters: AUC(0-inf), and Cmax Ratio: Test/Reference (Mesylate/HCI) | SAC [1] |

## 14.12.10. Pharmacokinetic Figures

| Pharma | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Bioavai | Bioavailability | | | | |
| 4.1. | PK | PK16b | Individual Plasma GSK3640254 Concentration-Time Plots (Linear and Semi-log) | Linear and Semi-Log Scale Paged by participant, overlay all treatments for each participant. Include LOQ line in plot. | SAC [1] |
| 4.2. | PK | PK17 | Mean Plasma GSK3640254 Concentration-Time Plots (Linear and Semi-log) | Linear and Semi-Log Scale By treatment. Use nominal times in X axis. | SAC [1] |
| 4.3. | PK | PK18 | Median Plasma GSK3640254 Concentration-Time Plots (Linear and Semi-log) | Linear and Semi-Log Scale By treatment. Use nominal times in X axis. | SAC [1] |
| 4.4. | PK | PK28 | Geometric Mean Treatment Ratio and 90% Confidence Interval of GSK3640254 PK Parameters for Relative Bioavailability | Ratio: Test/Reference<br>(Mesylate/HCI) | SAC [1] |
| 4.5. | PK | PK25 | Comparative Plot of Individual Plasma GSK3640254 PK Parameters for Relative Bioavailability by treatment (Linear and Semi-log) | | SAC [1] |

#### 14.12.11. Pharmacokinetic Population (PopPK) Tables

Not applicable.

### 14.12.12. Pharmacokinetic Population (PopPK) Figures

Not Applicable

#### 14.12.13. Pharmacodynamic Tables

Not applicable.

#### 14.12.14. Pharmacodynamic Figures

Not applicable.

### 14.12.15. Pharmacokinetic / Pharmacodynamic Tables

Not applicable.

#### 14.12.16. Pharmacokinetic / Pharmacodynamic Figures

Not applicable.

## 14.12.17. ICH Listings

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title Programming Note | | Deliverable<br>[Priority] |
| Subje | Subject Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC [1] |
| 2. | Safety | ES3 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC [1] |
| 3. | Safety | SD3 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC [1] |
| 4. | Safety | TA2 | Listing of Planned and Actual Treatments | IDSL | SAC [1] |
| Protoc | col Deviations | | | | |
| 5. | Safety | DV2A | Listing of Important Protocol Deviations | ICH E3 | SAC [1] |
| 6. | Safety | IE4 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC [1] |
| Popul | Populations Analysed | | | | |
| 7. | Safety | SP3A | Listing of Participants Excluded from Any Population | ICH E3 | SAC [1] |
| Demographic and Baseline Characteristics | | | | | |
| 8. | Safety | DM4 | Listing of Demographic Characteristics | ICH E3 | SAC [1] |
| 9. | Safety | DM10 | Listing of Race | ICH E3 | SAC [1] |
| Prior and Concomitant Medications | | | | | |
| 10. | Safety | CP_CM4 | Listing of Concomitant Medications | IDSL | SAC [1] |

| ICH: I | _istings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Expo | sure and Treat | ment Compli | ance | | |
| 11. | Safety | EX4 | isting of Exposure Data ICH E3 | | SAC [1] |
| 12. | Safety | Non-<br>Standard2 | Listing of Meal Data Identical to study 207187 Listing 54 | | SAC [1] |
| Adve | rse Events | | | | |
| 13. | Safety | AE9CP | Listing of All Adverse Events | ICH E3 | SAC [1] |
| 14. | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | ICH E3 | SAC [1] |
| 15. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | | SAC [1] |
| Serio | us and Other S | Significant A | dverse Events | | |
| 16. | Safety | AE9CPa | Listing of Serious Adverse Events | ICH E3 | SAC [1] |
| 17. | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | ICH E3 | SAC [1] |
| 18. | Safety | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | ICH E3 | SAC [1] |
| Hepat | tobiliary (Liver | ) | | | |
| 19. | Safety | MH2 | Listing of Medical Conditions for Participants with Liver Stopping Events | IDSL | SAC [1] |
| 20. | Safety | SU2 | Listing of Substance Use for Participants with Liver Stopping Events | IDSL | SAC [1] |
| 21. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | IDSL | SAC [1] |
| All La | boratory | | | | |
| 22. | Safety | LB13 | Listing of Reference Ranges for Clinical Laboratory Tests | | SAC [1] |
| 23. | Safety | LB6 | Listing of Clinical Chemistry Data | | SAC [1] |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title Programming Notes | | Deliverable<br>[Priority] |
| 24. | Safety | LB6 | Listing of Hematology Data | | SAC [1] |
| 25. | Safety | UR2B | Listing of Urinalysis Data | isting of Urinalysis Data | |
| 26. | Safety | LB6 | Listing of All Clinical Chemistry Laboratory Data for Participants with Any Value of Potential Clinical Importance OR Outside Normal Range | ICH E3. Display ALL labs for a subject who experienced a value of potential clinical importance or a value outside of normal range | SAC [1] |
| 27. | Safety | LB6 | Listing of Clinical Chemistry Laboratory Values of Potential Clinical Importance | | SAC [1] |
| 28. | Safety | LB6 | Listing of All Hematology Data for Participants with Any Value of Potential Clinical Importance OR Outside Normal Range | ICH E3. Display ALL labs for a subject who experienced a value of potential clinical importance or a value outside of normal range | SAC [1] |
| 29. | Safety | LB6 | Listing of Hematology Laboratory Values of Potential Clinical Importance | | SAC [1] |
| 30. | Safety | LB14 | Listing of Laboratory Data with Character Results | ICH E3 | SAC [1] |
| ECG | | | | | |
| 31. | Safety | EG4 | Listing of All ECG Findings | IDSL. Sort by treatment/period and visit | SAC [1] |
| 32. | Safety | EG6 | Listing of Abnormal ECG Findings | IDSL | SAC [1] |

| ICH: L | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 33. | Safety | EG4 | Listing of All ECG Values for Participants with Any Value of Potential Clinical Importance | IDSL. Display ALL ECGs for a subject who experienced a value of potential clinical importance Display ALL ECGs for a subject who experienced a value of potential clinical importance. | SAC [1] |
| Vital S | Vital Signs | | | | |
| 34. | Safety | VS5 | Listing of Vital Signs | IDSL | SAC [1] |
| 35. | Safety | VS5 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL. Display ALL vital signs for a subject who experienced a value of potential clinical importance | SAC [1] |

# 14.12.18. Non-ICH Listings

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Pharmacokinetic Statistical Analysis | | | | | |
| 36. | PK | SAS<br>output of<br>Table 4.4 | SAS Output of Summary Results of GSK3640254 PK Parameter Treatment Comparisons for the Relative Bioavailability | | SAC [1] |

## 14.13. Appendix 13: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request